CLINICAL TRIAL: NCT00363350
Title: Rituximab for the Treatment of Primary Sjögren's Syndrome: a Double Blinded Randomized Placebo-Controlled Trial
Brief Title: Rituximab Treatment in Sjogren's Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: H Bootsma, University Medical Centre Groningen
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: METc2005.229
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: rituximab (anti-CD20) — 2 infusions of 1000 mg
  Other Names: Mabthera

SUMMARY:
This study is an evaluation of the effect of rituximab compared to placebo in combination with steroids on salivary flow and serological and clinical parameters in patients with primary SS.

DETAILED DESCRIPTION:
Study design:

phase II trial

Study objective:

evaluation of the effect of rituximab compared to placebo in combination with steroids on salivary flow and serological and clinical parameters in patients with primary SS

Number of participating centres:

1

Duration:

follow-up 48 weeks

Study medication:

2 infusions on day 1 and day 15 rituximab infusions (1000 mg) or placebo infusions intravenous infusion of 100 mg of methylprednisolone before infusion of rituximab (or the placebo for rituximab), together with 60 mg per day of oral prednisone on days 2, 3, 16 and 17, 30 mg per day on days 4, 5, 18 and 19 and 15 mg per day on days 6 and 20

Primary objective/endpoint:

stimulated salivary gland function (stimulated submandibular/sublingual and parotid saliva)

Secondary objectives/endpoint:

Functional parameters Laboratory parameters Subjective parameters Histological/Molecular parameters

Number of subjects:

30 patients with primary SS (20 patients rituximab treatment, 10 patients placebo)

ELIGIBILITY:
Inclusion Criteria:

* Stimulated whole saliva secretion ≥ 0,15 ml/min
* Male or female > 18 years
* Primary SS according to the revised European - U.S. criteria(22)
* Positive autoantibodies (IgM-Rf > 10 and SS-A and/or SS-B)
* Parotid gland biopsy (paraffine material and fresh frozen tissue) with characteristic features of SS performed at time of inclusion (no longer than 12 months ago)
* Use of reliable method of contraception during the study
* Written informed consent

Exclusion Criteria:

* The presence of any other connective tissue disease
* Preceding treatment with anti-TNF or other monoclonal antibodies
* Use of prednisone, hydroxychloroquine less than 1 month ago
* Use of MTX, cyclophosphamide, cyclosporin, azathioprine and other DMARDS less than 0,5 year ago
* Serum creatine > 2.8 mg/dl (250 micromol/l)
* ASAT or ALAT outside 1.5 x upper normal range of the laboratory
* Hb < 9 g/dl (5.6 mmol/l) for males and 8.5 g/dl (5.3 mmol/l) for females
* Neutrophil granulocytes less than 0.5 x 109/l
* Platelet count less then 50 x 109/l
* Positive pregnancy test or breast-feeding
* History of alcohol or drug abuse
* Serious infections
* Underlying cardiac, pulmonary, metabolic, renal or gastrointestinal conditions, chronic or latent infectious diseases or immune deficiency which places the patient at an unacceptable risk for participation in the study
* History of any malignancy with the exception of completely resected basal cell carcinoma of the skin

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
stimulated whole salivary flow rate | 48 weeks

SECONDARY OUTCOMES:
Functional parameters | 48 weeks
Laboratory parameters | 48 weeks
Subjective parameters | 48 weeks
Histological/Molecular parameters | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jiska Meijer, MD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Background] Pijpe J, van Imhoff GW, Spijkervet FK, Roodenburg JL, Wolbink GJ, Mansour K, Vissink A, Kallenberg CG, Bootsma H. Rituximab treatment in patients with primary Sjogren's syndrome: an open-label phase II study. Arthritis Rheum. 2005 Sep;52(9):2740-50. doi: 10.1002/art.21260. PMID 16142737
- [Derived] Meijer JM, Meiners PM, Vissink A, Spijkervet FK, Abdulahad W, Kamminga N, Brouwer E, Kallenberg CG, Bootsma H. Effectiveness of rituximab treatment in primary Sjogren's syndrome: a randomized, double-blind, placebo-controlled trial. Arthritis Rheum. 2010 Apr;62(4):960-8. doi: 10.1002/art.27314. PMID 20131246